CLINICAL TRIAL: NCT04361058
Title: Graft-Versus-Tumor Augmentation With Nivolumab for High-Risk Patients With MDS and AML After Allogeneic Stem Cell Transplantation Using Post-Transplantation Cyclophosphamide
Brief Title: Nivolumab for High-Risk MDS/AML Patients After Allogeneic Stem Cell Transplant With Post-Transplant Cyclophosphamide
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The single site that was deemed appropriate for this study was unable to enroll patients. Closed due to slow accrual.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT 30; CA209-9WP (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2021-04

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myelodysplastic Syndrome Acute Myeloid Leukemia
Keywords: Graft versus host disease; Allogeneic stem cell transplant; Nivolumab; Myelodysplastic syndrome; Acute myeloid leukemia; Post-transplant cyclophosphamide
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; GATA2 Deficiency; Graft vs Host Disease | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - HLA-matched unrelated donor SCT treated with Nivolumab (Experimental): AML/MDS participants who have allogeneic stem cell transplants with an HLA-matched unrelated donor will be separated into Arm A and treated with Nivolumab post-SCT
  Interventions: Drug: Nivolumab
- Arm B - HLA-haploidentical donor SCT treated with Nivolumab (Experimental): AML/MDS participants who have allogeneic stem cell transplants with a HLA-haploidentical donor will be separated into Arm B and treated with Nivolumab post-SCT
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — At Day +50 (±10 days) post-allogeneic SCT, participants will be treated with Nivolumab. Nivolumab will be administered intravenously once every two weeks for a total of 4 treatments. Participants will initially receive nivolumab at a significantly reduced starting dose of 0.25 mg/kg. This dose was determined based on the incidence of increased aGVHD, which was noted after treatment post-SCT in previous studies. Nivolumab IV will be given every 2 weeks for 4 cycles. One dose of nivolumab is equivalent to one cycle. The first administration will be at Day +50 (±10 days), assuming the participant has not had any evidence of Grade II-IV aGVHD after allogeneic SCT and does not have any current evidence of any grade of aGVHD at the day of first application of nivolumab. Depending on emerging safety data, dose escalation cohorts will explore higher dose levels of nivolumab at 0.5 mg/kg and 1 mg/kg.
  Other Names: Opdivo

SUMMARY:
There are no strategies developed post-stem cell transplant (SCT) for patients who receive allogenic SCT with a significant amount of blasts prior SCT. Novel strategies to treat relapsed AML/MDS and to reduce the incidence of relapse after allogeneic SCT are needed. This study is being done in patients with high-risk MDS or AML who undergo an allogeneic SCT.

The study will have two arms, participants who receive an HLA-matched unrelated donor SCT (Arm A) or HLA- haploidentical SCT (Arm B). Following myeloablative conditioning (MAC), GVHD prophylaxis with post-transplantation cyclophosphamide (PTCy), tacrolimus and mycophenolate mofetil will be given per standard of care. At 40-60 days post SCT, If the patient has not had any evidence of Grade II-IV acute graft-versus-host-disease (aGVHD), Nivolumab will be given intravenously every 2 weeks for 4 cycles of consolidation or treatment with Nivolumab. Dose-escalation of Nivolumab will follow the standard 3+3 design where a maximum of three dose levels will be evaluated, with a maximum of 18 patients treated with nivolumab per arm. As the maximum tolerated dose (MTD) of Nivolumab may differ between Arm A and Arm B, dose escalation of nivolumab in each arm will be followed separately following allogeneic SCT. Immunosuppression with tacrolimus will be continued during the cycles of PD-1 blockade to provide a moderate level of GVHD prophylaxis during consolidation or treatment with nivolumab.

DETAILED DESCRIPTION:
There are no strategies developed post SCT for patients who receive allogenic SCT with a significant amount of blasts prior SCT. Historically, the risk of relapse for patients with high-risk myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) is estimated to be 60% to 80%. No standard consolidation treatment options for patients with AML/MDS have been established to decrease the risk of relapse. The options are also limited for patients with relapsed disease after allogeneic SCT. Thus, novel strategies to treat relapsed disease and to reduce the incidence of relapse after allogeneic SCT are needed. PD-1 inhibition can induce remission in patients with relapsed hematologic disease after allogeneic SCT, but the major risk of PD-1 blockade after allogeneic SCT remains the promotion of severe GVHD leading to death. Alternative approaches are needed to reduce the incidence of GVHD after PD-1 blockade while maintaining a strong graft-versus-tumor (GVT) effect. Adding post-transplantation cyclophosphamide (PTCy) prior to PD-1 blockade after an allogeneic SCT may potentially reduce the expected incidence of acute GVHD and prevent relapse by enhancing the GVT effect. As the absence of GVHD has been associated with increased incidence of relapse, it is reasonable to investigate high-risk patients in CR without evidence of GVHD after allogeneic SCT. Since early relapse or progression of disease after allogeneic SCT is associated with a very poor outcome and treatment options are limited, it is also reasonable investigate patients with persistent or progressive disease after allogeneic SCT. At present, no prospective studies have been conducted post-allogeneic SCT using PTCy followed by PD-1 inhibition as a consolidation therapy or as a therapy for persistent or progressive disease. PD-1 blockade after PTCy appears to be safe and does not induce GVHD when compared to patients who did not receive PD-1 blockade after PTCy. As a means to reduce the risk of relapse or provide potentially effective treatment for persistent/progressive disease, this strategy may also avoid the harm of inducing GVHD or possibly exacerbating previously existing GVHD.

This is a multi-center, open-label, double-arm Phase I dose-escalation study of patients with high-risk MDS and AML prior to receiving allogeneic SCT. A maximum of 36 patients (maximum 18 patients per arm) are planned to be screened and enrolled prior to allogeneic SCT with the expectation that each patient will be a suitable candidate for study participation at the time of administration of nivolumab.

Following myeloablative conditioning (MAC) and HLA-matched unrelated donor SCT (Arm A) or HLA- haploidentical SCT (Arm B), GVHD prophylaxis with PTCy, tacrolimus and mycophenolate mofetil will be given per standard of care.

At 40-60 days post SCT, patients without evidence of aGVHD will begin 4 cycles of consolidation or treatment with nivolumab. Immunosuppression with tacrolimus will be continued during the cycles of PD-1 blockade to provide a moderate level of GVHD prophylaxis during consolidation or treatment with nivolumab.

As the maximum tolerated dose (MTD) of nivolumab may differ between Arm A and Arm B, dose escalation of nivolumab in each arm will be followed separately following allogeneic SCT. Dose-escalation of Nivolumab will follow the standard 3+3 design where a maximum of three dose levels will be evaluated, with a maximum of 18 patients treated with nivolumab per arm. Nivolumab IV will be given every 2 weeks for 4 cycles. One dose of nivolumab is equivalent to one cycle. The first administration will be at Day +50 (±10 days), assuming the patient has not had any evidence of Grade II-IV aGVHD after allogeneic SCT and does not have any current evidence of any grade of aGVHD at the day of first application of nivolumab.

Participants will be followed for up to 1 year post-SCT and have long-term follow-up will be from 1.5 up to 3 years post-SCT for adverse events, progression or relapse, survival, and evidence of GVHD.

Chronic GVHD staging and grading will be assessed for efficacy as per National Institutes of Health Consensus criteria. Safety and tolerability will be assessed as per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03.

ELIGIBILITY:
Inclusion Criteria for initial enrollment:

* Written informed consent form (ICF), according to local guidelines, signed by the patient or by a legal guardian prior to the performance of any study-related screening procedures (i.e., prior to conditioning).
* Male and female patients between ≥18 and ˂66 years-of-age
* Patients with high-risk AML defined as: AML with ≥5% bone marrow blast burden prior to allogeneic SCT who failed ≥2 lines of cytoreductive anti-leukemic therapy
* Patients with high risk MDS defined as: MDS with ≥10% bone marrow blasts prior to allogeneic SCT despite 1 line of prior cytoreductive anti-leukemic treatment with chemotherapy or hypomethylating agent
* Patients will receive a MAC MUD or MAC haploidentical SCT followed by PTCy as treatment for AML or MDS.
* A 10/10 HLA-match is required for patients that will receive a MUD SCT.
* A 5/10 HLA-match or greater is required for patients that will receive a haploidentical SCT.
* Patients must be able to swallow and retain oral medication.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or

Inclusion Criteria after SCT, prior to start of nivolumab:

* Patients who have achieved a CR post-allogeneic SCT
* Patients who have persistent disease post-allogeneic SCT
* Greater than 50% PB donor T cell chimerism
* Adequate renal function defined as serum creatinine ≤2.0 mg/dL or creatinine clearance ≥40 mL/min measured or calculated by Cockcroft-Gault equation.
* Females of childbearing potential must have a negative serum or urine pregnancy test result within 72 hours prior to the first dose of nivolumab and must agree to follow instructions for method(s) of contraception, using two forms of acceptable contraception, including one barrier method, for the duration of treatment with nivolumab and for 7 months following their last dose of the study drug. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy.
* Male patients with female partners of childbearing potential are required to use contraceptive methods, during their participation in the study and for 7 months following the last dose of study drug. Male patients must also refrain from donating sperm during their participation in the study and for 7 months following the last dose of study drug.
* Ability to understand the nature of this study and to comply with study and follow-up procedures.

Exclusion Criteria for initial enrollment:

* Prior allogeneic SCT
* Pregnant or lactating women
* Evidence of active uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of active infection progression are present. This is assessed by the site clinicians including consulting physicians from infectious disease regarding adequacy of therapy. These infections include, but are not limited to:

  * Known human immunodeficiency virus (HIV) infection
  * Active tuberculosis infection
* History of autoimmune pneumonitis within the last 5 years
* Prior diagnosis of an inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of severe hypersensitivity reactions to monoclonal antibodies
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Exclusion Criteria after SCT, prior to start of nivolumab:

* Current evidence of any grade of active aGVHD at Day 40-60 at the time of study enrollment
* Prior history of Grade II or higher aGVHD (Appendix E)
* Prior or concurrent treatment with DLI
* Use of a study drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of nivolumab, except antimicrobial drugs. For study drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the study drug and administration of nivolumab is required, except antimicrobial drugs.
* Evidence of active uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of infection progression are present.
* Active autoimmune disease that has persisted or recurred after allogeneic SCT, except vitiligo or resolved childhood asthma/atopy.
* Inadequate organ function:

  * Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months of enrollment, New York Heart Association Class III or IV congestive heart failure (Appendix B), circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy. If the patient does not meet the minimum criteria and/or receive cardiotoxic agents, cardiology consultation and clearance is recommended.
  * Significant respiratory disease that requires mechanical ventilation support or a resting O2 saturation <90% by pulse oximetry. FEV1/FVC/DLCO <50%. If the patient does not meet the minimum criteria, pulmonary consultation and clearance is recommended.
  * Serum creatinine ≥2.0 mg/dL. If the patient does not meet the minimum criteria, nephrology consultation and clearance is recommended.
  * Serum bilirubin >2.5 mg/dL (except for hemolysis or Gilbert's syndrome) and transaminases ≥3 upper limit of normal (ULN). If the patient does not meet minimum criteria, hepatology consultation and clearance should be considered. If warranted, a liver biopsy should be performed prior to transplant.
* Any corticosteroid therapy for indications other than GVHD at doses >1 mg/kg/day methylprednisolone or equivalent within 7 days of start of nivolumab.
* Any corticosteroid therapy for prior GVHD including topicals, budesonide and beclomethasone PO at any dose within 7 days of start of nivolumab.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities as a determinant of the Maximum Tolerated Dose (MTD) | After the first dose of Nivolumab treatment for up to 28 days.
  Defined as the highest dose at which ≤ 1 of 6 participants experience a DLT. Certain toxicities will be considered dose-limiting unless clearly attributable to an extraneous cause, such as underlying disease. If 2 or more patients in a dosing group of ≤6 patients experience a DLT, the MTD has been exceeded. If 2 or more patients in a dosing group of up to 6 patients experience a DLT and only 3 patients were evaluated at the previous dose (i.e. next lower). Then, an additional 3 patients will be evaluated at this next lower dose, and if zero or one have DLTs, then this previous dose level is declared the MTD. Dose level -1 will be tested if dose level 1 exceeds the MTD.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | PFS will be assessed for up to 3 years post-SCT
  Defined as the time from the first day of study drug administration until the date of relapse, progression, or death from any cause; patients not known to have relapsed/progressed or died at last follow-up are censored on the date they were last examined. Progression is defined as evidence for an increase in bone marrow blast percentage and/or increase of absolute blast counts in the blood: >50% increase in marrow blasts over baseline (min 15% increase is required in cases with <30% blasts at baseline); or persistent marrow blast percentage of >70% over at least 3 months; without at least a 100% improvement in absolute neutrophil count (ANC) to an absolute level [>0.5 x 109/L (500/μL), and/or platelet count to >50 x 109/L (50,000/μL) non-transfused]; or >50% increase in peripheral blasts (WBC x % blasts) to >25 x 109/L (>25,000/μl) (in the absence of differentiation syndrome); or New extramedullary disease.
Overall survival (OS) | OS will be assessed for up to 3 years post-SCT
  Defined as the time from the first day of study drug administration to death on study from any cause or study discontinuation.
Number of participants that experience Non-relapse mortality | Will be assessed throughout study treatment, when study treatment ends, and for up to 3 years
  Defined as death in the absence of recurrent or progressive malignancy after stem cell transplant (SCT).
Number of participants with evidenceof cGVHD | Will be assessed throughout study treatment, when study treatment ends, and for up to 3 years
  Number of participants with evidence/cumulative incidence of chronic GVHD (>0 cGVHD symptoms on the chronic GVHD activity assessment form) at 1 year and up to 3 years post-SCT.
Number of participants that experience Nivolumab-related mortality | Will be assessed throughout study treatment, when study treatment ends, and for up to 3 years
  Number of participants with mortality directly related to nivolumab leading to Grade III-IV aGVHD or non-GVHD immune-mediated toxicity leading to death.
Number of participants who relapse (CIR) | Will be assessed throughout study treatment, when study treatment ends, and for up to 3 years
  Number of participants (cumulative incidence) who achieve a complete remission (CR) or CR with incomplete hematologic recovery (CRi) who later relapse (Bone marrow blasts ≥5%; or reappearance of blasts in the blood; or development of extramedullary disease) measured from the date of achievement of a remission until the date of relapse.
Relapse free survival (RFS) | Will be assessed for up to 3 years
  Defined as the time measured from the date of achievement of a remission until the date of relapse (bone marrow blasts ≥5%; or reappearance of blasts in the blood; or development of extramedullary disease) or death from any cause; only for patients achieving complete remission (CR), or CR with incomplete hematologic recovery (CRi); patients not known to have relapsed or died at last follow-up are censored on the date they were last examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado Blood Cancer Institute, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No